CLINICAL TRIAL: NCT01756027
Title: Feasibility Study: Evaluation of the Effectiveness and Safety of the Ulthera® System for Treatment of Erythematotelangiectatic Rosacea
Brief Title: Feasibility Study: Ulthera System for the Treatment of Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULT-131
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-11

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: Rosacea; Ulthera System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for the skin
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Ulthera System providing one treatment per cheek
  Interventions: Device: Ulthera System providing one treatment per cheek
- Group B (Active Comparator): Ulthera System providing two treatments per cheek
  Interventions: Device: Ulthera System providing two treatments per cheek

INTERVENTIONS:
Device: Ulthera System providing one treatment per cheek — Focused ultrasound energy delivered below the surface of the skin per cheek.
  Other Names: Ultherapy™
  Arms: Group A
Device: Ulthera System providing two treatments per cheek — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™
  Arms: Group B

SUMMARY:
Up to 12 subjects will be enrolled. Enrolled subjects will receive one or two Ultherapy treatments on the cheeks, depending on their assigned study group. Follow-up visits will occur 14, 30 and 90 days post-treatment. Study images will be obtained pre-treatment, 30-60 min post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This study is a prospective, randomized, single-center clinical trial. The study will be conducted in two Phases. In Phase I, subjects will be assigned to one of two treatment groups. One study group will receive one dual depth Ultherapy treatment to a region on the cheeks, and one study group will receive two dual depth Ultherapy treatments to a region on the cheeks 14 days apart. Average pain scores will be obtained using a Numeric Rating Scale following each region of treatment and for each depth of treatment. In Phase II, based on observations of last follow-up visit in Phase I (at 90 days after treatment), subjects will be given the option to receive treatment of the affected area(s) for the protocol specified region, treated at the treatment depth showing the most efficacy in Phase I. Efficacy will be determined by improvement in Erythematotelangiectatic Rosacea in the treatment area versus control (an untreated area) as determined by primary investigator assessment at the last follow-up visit in Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years.
* Subject in good health.
* Clinical diagnosis of Erythematotelangiectatic Rosacea.
* Understands and accepts the obligation not to undergo any other procedures in the area(s) to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography and adherence to photography requirements.
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1.

Exclusion Criteria:

* Presence of an active systemic disease that may affect wound healing.
* Prominent telangiectases in the area(s) to be treated.
* History of post-inflammatory hyperpigmentation.
* Papulopustular or Phymatous Rosacea.
* Severe solar elastosis.
* Significant scarring in area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Presence of a metal stent or implant in the area(s) to be treated.
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatments to the intended treatment area(s) within six weeks prior to study participation or during the study.
* Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation,noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* History of the following cosmetic treatments in the area(s) to be treated:

  1. Skin tightening procedure within the past year;
  2. Injectable filler of any type within the past:

     * 12 months for Hyaluronic acid fillers (e.g.,Restylane)
     * 12 months for Ca Hydroxyapatite fillers (e.g., Radiesse)
     * 24 months for Poly-L-Lactic acid fillers (e.g., Sculptra)
     * Ever for permanent fillers (e.g., Silicone, ArteFill)
  3. Neurotoxins within the past three months;
  4. Ablative resurfacing laser treatment;
  5. Nonablative, rejuvenative laser or light treatment within the past six months;
  6. Surgical dermabrasion or deep facial peels
* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Topical Retinoids within the past two weeks;
  3. Antiplatelet agents / Anticoagulants (Coumadin, Heparin, Plavix);
  4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Improvement in Erythematotelangiectatic Rosacea of treatment area versus control | 90-days post-treatment treatment
  As determined by Primary Investigator assessment

SECONDARY OUTCOMES:
Improvement in Erythematotelangiectatic Rosacea of treatment area versus control (untreated area) | Participants will be followed for 90-days post treatment #1 (Group A) or post-treatment #2 (Group B)
  As determined by a live patient assessment and investigator designation of improved versus not improved for the area treated compared to the surrounding area at follow-up in Phase I

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lupin, M.D., Principal Investigator — Cosmedica
Locations (1):
- Cosmedica, Victoria, British Columbia, Canada